CLINICAL TRIAL: NCT05224375
Title: A Trial Evaluating the Safety and Effectiveness of the Laminar Left Atrial Appendage Closure System in Subjects With Non-Valvular Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laminar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-0039
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Closure of the left atrial appendage with the Laminar Left Atrial Appendage Closure system.
  Interventions: Device: Left Atrial Appendage Closure

INTERVENTIONS:
Device: Left Atrial Appendage Closure — Closure of the left atrial appendage with the Laminar Left Atrial Appendage Closure System

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Laminar Left Atrial Appendage Closure System to treat patients with non-valvular atrial fibrillation that cannot take, or a have a reason to seek an alternative to anticoagulant medications.

DETAILED DESCRIPTION:
Left atrial appendage closure (LAAC) is an approved therapy for stroke prevention in atrial fibrillation patients who are recommended for chronic oral anticoagulation therapy (OAC), but are non-eligible or have an appropriate rationale to seek a non-pharmacologic alternative to chronic oral anticoagulants in accordance with evidence-based decision-making criteria and current scientific guidelines.

The objective of this study is to evaluate the safety and effectiveness of the Laminar Left Atrial Appendage Closure System to treat patients with non-valvular atrial fibrillation who are deemed appropriate for LAAC to reduce the risk of stroke and systemic embolism.

Patients will be followed for 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with documented Non-Valvular AF, defined as AF (paroxysmal, persistent, or permanent) in the absence of moderate-to-severe mitral stenosis or a mechanical heart valve.
2. Subject must be ≥18 years of age.
3. Subject has a calculated CHA2DS2-VASc score of 2 or greater, denoting a high risk for stroke or systemic embolism.
4. Subject is recommended for chronic oral anticoagulation therapy (OAC), but is non eligible or has an appropriate rationale to seek a non-pharmacologic alternative to chronic OAC
5. Subject deemed appropriate for LAA closure by the Site Heart Team
6. Subject is eligible for the post-procedural antithrombotic regimen per protocol
7. Subject (or legally authorized representative, (where allowed)) has been informed of the nature of the study, agrees to its provisions, is willing and able to comply with the protocol-required medications and follow-up visits, and has provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Exclusion Criteria:

1. AF single episode or transient or reversible (e.g., secondary thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
2. Recent (within 90 days pre-procedure) stroke or transient ischemic attack
3. Subject with history of acute or recent myocardial infarction (MI) or unstable angina within 90 days
4. Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2, or dialysis at the time of screening
5. Active infection with bacteremia
6. Active COVID-19 infection
7. Cardiac tumor
8. Subject with a history of pericarditis, rheumatic heart disease, or severe cardiac valvular disease
9. Medical condition (other than AF) that mandates chronic oral anticoagulation (e.g., history of unprovoked deep vein thrombosis or pulmonary embolism, or mechanical heart valve)
10. Severe heart failure (New York Heart Association Class III or IV)
11. Documented symptomatic carotid artery disease (>50% diameter stenosis with prior ipsilateral stroke or TIA) or known asymptomatic carotid artery disease (diameter stenosis of >70%)
12. Prior cardiac surgery, history of mitral valve replacement or transcatheter mitral valve intervention, or any mechanical valve implant
13. Previous AF Ablation procedure in the 90 days before the LAMINAR procedure date
14. Need for AF Ablation procedure to be performed less than 90 days from the LAMINAR procedure
15. Subject with a history of coronary artery bypass graft (CABG) surgery
16. Recent (within 30 days pre-procedure) or planned (within 60 days postprocedure) cardiac or non-cardiac interventional or surgical procedure
17. Intracardiac thrombus or dense spontaneous echo contrast, as visualized by TEE within 2 days prior to implant
18. Left ventricular ejection fraction (LVEF) <30%
19. Circumferential pericardial effusion >10 mm or symptomatic pericardial effusion, signs or symptoms of acute or chronic pericarditis, or evidence of tamponade physiology
20. Atrial septal defect that warrants closure
21. High risk patent foramen ovale (PFO), defined as an atrial septal aneurysm (exclusion >15 mm or length > 15 mm) or large shunt (early [within 3 beats] or substantial passage of bubbles)
22. Moderate or severe mitral valve stenosis (mitral valve area <1.5 cm2)
23. Complex atheroma with mobile plaque of the aorta
24. Anatomic conditions that would prevent performance of a LAA occlusion procedure (e.g., prior atrial septal defect (ASD) or patent foramen ovale (PFO) surgical repair or implanted closure device, or obliterated or ligated left atrial appendage).
25. Vascular access precluding delivery of implant with catheter-based system
26. Subject with inferior vena cava (IVC) filter that would interfere with Laminar sheath insertion
27. Patient is unable to undergo general anesthesia
28. Patient has a condition which precludes adequate transesophageal echocardiographic (TEE) assessment
29. Patient has a known allergy, hypersensitivity or contraindication to aspirin, heparin, or device materials (e.g., nickel, titanium, gold) or that would preclude any P2Y12 inhibitor therapy (e.g., clopidogrel, ticlopidine, ticagrelor, prasugrel)
30. The patient has contrast sensitivity that cannot be adequately premedicated
31. Bleeding diathesis or coagulopathy
32. Thrombocytopenia (platelet count <75,000 cells/mm3), thrombocytosis (>700,000 cells/mm3), or leukopenia (white blood cell count <3,000 cells/mm3)
33. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following the index procedure. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to index procedure.
34. Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol or protocol-specified medication regimen, confound the data interpretation, or is associated with a life expectancy of less than 2 years
35. Current participation in another investigational drug or device study
36. Vulnerable Patients groups (minors, cognitively impaired persons, prisoners, persons whose willingness to volunteer could be unduly influenced by the expectation of benefits associated with participation or of refusal to participate, such as students, residents, and employees)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Closure success using the Laminar Left Atrial Appendage Closure System | 45 days
  Confirmation of functional LAA closure as defined by absence of residual peri-device flow ≤ 5mm in width per transesophageal echocardiography.
Adverse Events | 7 days and 45 days
  Rate of all cause-mortality and major adverse events (including procedure-related stroke, systemic embolism, life-threatening or major bleeding) and device- or procedure-related events requiring open cardiac surgery or major endovascular intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No